CLINICAL TRIAL: NCT05506475
Title: Evaluation of HCV Care and Treatment for HIV-HCV Co-infected Patients in Decentralised Areas in Vietnam
Acronym: MOVIDA-Hep2
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-084
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: HIV Infection; Hepatitis C Infection
Keywords: Direct Acting Antiviral; Dried Blood Spots
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — DBS and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood samples — venous blood collected in a 5 mL EDTA tube

SUMMARY:
With the advent of direct acting antiviral (DAA) treatment in 2013, HCV elimination has become feasible. Still, achieving HCV elimination in resource-limited countries appears to be arduous as several challenges need to be addressed.

In remote settings, absence of HCV VL testing to identify those who require DAA and to monitor DAA success is a first issue. As of today, HCV VL testing is still restricted to central facilities in major cities. Blood sampling using DBS is an appealing option to allow HCV VL monitoring in remote settings as this option is inexpensive, does not require a cold chain for storage and transportation of the samples and can be implemented rapidly.

A second issue is DAA access that remains scarce due to logistical and financial limitations. However, more affordable generic DAA, some of them being WHO pre-qualified, are now available.

Vietnam is amongst the 20 countries with the highest HCV burden with an estimate of 1.5 million chronic HCV-infected people (HCV prevalence: 1.1%). As observed in many other settings, HCV prevalence is higher among vulnerable populations such as HIV-infected individuals and people who inject drugs (PWID).

Vietnam has the will to increase access to DAA in the whole country. However, in remote settings, only some clinical sites will be allowed to dispense DAA. Discussions with the MoH of Vietnam brought to our knowledge that not all clinical sites caring for HIV patients and providing ART will dispense DAA.

Thus, some HIV-HCV co-infected patients will be followed in clinical sites where they will receive both antiretroviral therapy and DAA, while some other patients will continue to be followed for HIV in their usual clinical site but will be asked to visit another clinical site for HCV care and to receive DAA. We anticipate that the proportion of patients who will comply with the 12-week DAA will be lower in patients followed for HIV and HCV in two clinical sites than in those followed in a single clinical site.

DETAILED DESCRIPTION:
In 2015, it was estimated that 71 million people were chronically infected with hepatitis C virus (HCV) worldwide and that HCV accounted for a total of 1.34 million deaths, more than the number of deaths due to HIV. With the advent of direct acting antivirals (DAA) in 2013, HCV elimination has however become feasible. DAA treatment is essentially a combination of two DAA drugs from two different classes, having distinct mode of action against HCV. The rate of HCV cure after 12-week DAA treatment is usually >90%, whatever the genotype and even in presence of HIV co-infection. These very encouraging results led the WHO to launch the "elimination of viral hepatitis as a public health threat by 2030" acting plan, which targets, for HCV and hepatitis B virus (HBV), an overall 65% reduction in mortality and a 90% reduction in the number of new infections by 2030, as compared to the situation in 2015.

However, achieving HCV elimination in resource-limited countries appears to be arduous as several challenges still need to be addressed. HCV diagnosis is the first difficulty to overcome, but rapid diagnostic tests (RDT) which have largely been evaluated and present high sensitivity and specificity fulfilling standards of use allow to overcome this difficulty. Other barriers in the cascade of HCV care in remote settings include absence of HCV viral load (VL) testing to identify those who require DAA and to monitor DAA treatment success. As of today, HCV VL testing is still restricted to central facilities in major cities. Blood sampling using dried blood spots (DBS) is an appealing option to allow HCV VL monitoring in remote settings as this option is inexpensive, does not require a cold chain for storage and transportation of the samples and can be implemented rapidly. Moreover, DBS have been shown to perform well for HCV VL testing. Finally, DAA access remains scarce due to logistical and financial limitations. However, more affordable generic DAA, some of them being WHO pre-qualified, are now available.

Vietnam is amongst the 20 countries with the highest burden of HCV with an estimate of 1.5 million chronic HCV-infected people (HCV prevalence: 1.1%). Circulating HCV viruses are mainly genotype 1 and 6, subtypes 1a and 1b being the most common followed by 6a. As observed in many other settings, HCV prevalence is higher among vulnerable populations such as HIV-infected individuals (22.9% to 89.0%) and people who inject drugs (PWID) (74.0% to 87.0%). Moreover, PWID are core-transmitters with higher risk of re-infection than in the general population, which could compromise HCV eradication; a high rate of re-infection was found in PWID in Spain (9.8/100 PY) and in Bangladesh (4.2/100 PY).

Situation in Vietnam:

Vietnam has the will to increase access to HCV care in order to reach the World Health Organization (WHO) goals by 2030. As of today, DAA are almost exclusively available in national hospitals in large cities (i.e. Hanoi and Ho Chi Minh City). Its dispensation in remote settings is underway, but only a limited number of clinical sites will be selected to dispense DAA. Importantly, discussions with the Ministry of Health (MoH) of Vietnam brought to our knowledge that not all clinical sites caring for HIV patients will dispense DAA.

This means that, in remote settings, some HIV-HCV co-infected patients will be followed in one clinical site for both infections, while some other patients will be followed in one clinical site for HIV, and will be invited to visit another clinical site to receive DAA. This puts the latter at higher risk of DAA refusal and discontinuation.

Hence,Study Principal Investigators aim at comparing, in remote settings, in HIV-HCV co-infected patients, compliance with the 12-week DAA treatment between i) patients followed in the same clinical site for their HIV and HCV infections, and ii) patients followed in two clinical sites for their HIV and HCV infections.

To identify those who require DAA and monitor DAA treatment success, HCV VL testing is required. Yet, laboratories able to measure HCV VL are still scarce, limited to central level and no blood sample transfer network is currently implemented. Interventions to increase access to HCV VL testing are thus required. Point-of-care (POC) devices have been developed for HCV VL testing, but are not yet available in the field in Vietnam and costs, among other things, make that not all clinical sites could be equipped with them. An attractive option to rapidly scale-up HCV VL testing relies on the use of DBS as proposed by the WHO. Indeed, DBS facilitate sample transfer to a central laboratory and reduce the associated costs. Within this project, DBS use will be implemented for HCV VL testing.

The MOVIDA (Monitoring Of Viral load In Decentralised Area) Hep 2 project is therefore the opportunity to implement an intervention to increase HCV VL testing to support decentralisation of DAA access. This project will also provide valuable information to consolidate, adapt and expand the national programme against HCV in Vietnam, and will guide other resource-limited countries in the implementation of their own programmes against HCV.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrolment ≥18 years.
* Documented HIV-1 infection.
* HCV infection documented by the presence of Anti-HCV antibodies or a positive RDT; if the result was negative but dates from more than 6 months the patient will be tested again.
* Consent to participate in the study

Exclusion Criteria:

* HCV negative patient.
* Patient not routinely followed for HIV care in the clinical sites participating in the study.
* Previous treatment by DAA.
* Patient for whom the health status, according to the medical staff, may interfere with the study or is not compatible with the sampling planned in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-HCV co-infected adults already enrolled in HIV care
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
To compare compliance to the 12-week DAA treatment between patients followed in the same clinical site for HIV and HCV infections, and patients followed in two clinical sites for these two infections | 12 weeks
  Proportion of patients who have taken ≥90% of daily doses during the 12-week DAA (measured by pill count).

SECONDARY OUTCOMES:
To describe the compliance to the 12-week DAA treatment, and identify factors associated with good compliance | 12 weeks
  Number of days the DAA treatment was taken (measured by pill count),
To evaluate and compare the efficacy of the DAA treatment (defined by SVR12), and identify factors associated with SVR12 | 24 weeks
  Proportions of patients achieving SVR12, defined by an undetectable HCV VL 12 weeks after the planned end date of DAA treatment,
To describe the HCV genotypes circulating | 24 weeks
  Characterization of HCV genotypes and subtypes by means of Sanger sequencing
To describe HCV drug resistances in those not achieving SVR12, | 24 weeks
  Full-length HCV genome sequence analysis, by means of shotgun metagenomics using deep sequencing, for patients who did not achieve SVR12
To estimate the rate of HCV re-infection within 24 months after SVR12 | 30 months
  HCV VL measured 12 and 24 months after SVR12
To evaluate and compare quality of life in HIV-HCV co-infected patients before and after DAA treatment. | 18 months
  Quality of life evaluated through the 5-level EQ-5D version (EQ-5D-5L) quality of life scale (scale is numbered from 0 to 100, 100 means the best health the participant can imagine / 0 means the worst health the participant can imagine), measured prior to and 1 year after the end of DAA treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yoann MADEC, PhD, Principal Investigator — Institut Pasteur; Tuan Anh NGUYEN, PhD, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam; Thang Hong PHAM, PhD, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (2):
- Vietnam (2):
  - Center for Diseases Control and Prevention of Nghe An province, Vinh, Nghệ An Province
  - Center for Disease Control and Prevention of Yen Bai Province, Yên Bái, Yen Bai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran TH, Nguyen BT, Nguyen TA, Pham TTP, Nguyen TTT, Mai HTB, Pham HB, Nguyen TM, Phan HTT, Do NT, Ait-Ahmed M, Taieb F, Madec Y. Dried blood spots perform well to identify patients with active HCV infection in Vietnam. J Viral Hepat. 2020 May;27(5):514-519. doi: 10.1111/jvh.13263. Epub 2020 Feb 11. PMID 31981287